CLINICAL TRIAL: NCT01053065
Title: The Multicenter Atorvastatin Plaque Stabilization (MAPS) Study
Acronym: MAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Biomedical Foundation for Cardiovascular Research of Padova (Unknown); Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MAPS
Record Dates: First submitted 2010-01-20; First posted 2010-01-21 (Estimated); Last update posted 2021-04-30 (Actual); Status verified 2005-01

CONDITIONS: Symptomatic Carotid Stenosis; Hypercholesterolemia; Indication for Carotid Endarterectomy
Keywords: Atherosclerosis; Macrophages; Carotid arteries; Statin
MeSH Terms: conditions — Hypercholesterolemia; Atherosclerosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Atorvastatin 10 mg/day (Active Comparator): Arm composed of 20 patients, receiving atorvastatin 10 mg/day
  Interventions: Drug: Atorvastatin - Cholestyramine - Sitosterol
- Atorvastatin 80 mg/day (Active Comparator): Arm composed of 20 patients, receiving atorvastatin 80 mg/day
  Interventions: Drug: Atorvastatin - Cholestyramine - Sitosterol
- Cholestyramine - Sitosterol (Active Comparator): Arm composed of 20 patients receiving cholestyramine 8 g/day plus sitosterol 2.5 g/day
  Interventions: Drug: Atorvastatin - Cholestyramine - Sitosterol

INTERVENTIONS:
Drug: Atorvastatin - Cholestyramine - Sitosterol

SUMMARY:
The impact on cardiovascular events achieved by statin therapy seems to be mostly attributable to the cholesterol-lowering effect with a highly debated contribution of the lipid-independent pleiotropic effects. However, a short-term benefit has been documented for patients treated with statins in acute coronary syndromes and other clinical settings. These observations strengthened the hypothesis of additional, so-called pleiotropic actions of statins.

The investigators therefore sought to investigate how different lipid-lowering strategies (non-statin therapy, low-dose statin and high-dose statin) affects cellular composition of carotid plaque over a short-term period of three months. Specifically the investigators tried and dissect the LDL-C lowering impact on plaque cellular composition as compared to the lipid-independent contribution on plaque macrophage and smooth muscle cells.

DETAILED DESCRIPTION:
Patients (with Total Cholesterol (TC) ranging between 5.83-7.64 mmol/l), never treated with lipid lowering drugs, with symptomatic carotid stenosis >70% (NASCET criteria), and therefore eligible for carotid endarterectomy, were recruited. All patients were enrolled within 30 days from the clinical event, and randomized to one of three treatment groups. Each group, composed of 20 patients, received atorvastatin 10 mg/day (AT-10 group), or atorvastatin 80 mg/day (AT-80 group), or cholestyramine (Questran, Bristol Myer Squibb) 8 g/day plus sitosterol (Unilever) 2.5 g/day (C-S group) for three months prior to the vascular procedure. A placebo group was not included for ethical reasons due to the high cardiovascular risk profile in this population.

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic carotid stenosis > 70% (NASCET criteria)
* Eligibility for carotid endarterectomy
* Total cholesterol level between 5.83 and 7.64 mmol/L
* Never treated with lipid lowering drugs

Exclusion Criteria:

* Previous lipid lowering therapy
* Total cholesterol <5.83 or >7.64 mmol/L
* Evidence of chronic inflammatory disease (clinical and laboratory).
* Patients at high risk for cerebrovascular events (i.e. ulcerated carotid plaque, recurrent TIAs).

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)

PRIMARY OUTCOMES:
Changes in cellular composition of carotid plaque. | Three months

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pauletto, MD, Principal Investigator — University of Padova - Italy
Locations (3):
- Italy (3):
  - University of Chieti Medical School, Chieti
  - University of Padova Medical School, Padua
  - University of Padova Medical School - Treviso Branch, Treviso

REFERENCES:
- [Background] Pauletto P, Puato M, Faggin E, Santipolo N, Pagliara V, Zoleo M, Deriu GP, Grego F, Plebani M, Sartore S, Bon GB, Heymes C, Samuel JL, Pessina AC. Specific cellular features of atheroma associated with development of neointima after carotid endarterectomy: the carotid atherosclerosis and restenosis study. Circulation. 2000 Aug 15;102(7):771-8. doi: 10.1161/01.cir.102.7.771. PMID 10942746
- [Background] Faggin E, Zambon A, Puato M, Deeb SS, Bertocco S, Sartore S, Crepaldi G, Pessina AC, Pauletto P. Association between the --514 C-->T polymorphism of the hepatic lipase gene promoter and unstable carotid plaque in patients with severe carotid artery stenosis. J Am Coll Cardiol. 2002 Sep 18;40(6):1059-66. doi: 10.1016/s0735-1097(02)02116-2. PMID 12354428